CLINICAL TRIAL: NCT02724345
Title: The Effect of Postoperative Adjuvant TACE Treatment in CK18 Positive Patients of Hepatocellular Carcinoma.
Brief Title: Postoperative Adjuvant TACE Treatment in CK18 Positive Patients
Status: Completed | Type: Observational
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospital, Eastern Hepatobiliary Surgery Hospital
Other Study IDs: ZD201206002-P1
Record Dates: First submitted 2016-03-28; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Adjuvant TACE; Hepatocellular Carcinoma.
Keywords: Cell keratin 18
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CK18 positive: HCC patients with CK18 high expression levels in tumor tissue.
- CK18 negative: HCC patients with CK18 high expression levels in tumor tissue.

SUMMARY:
To evaluate and analyse the clinical effect and application value of postoperative adjuvant TACE treatment in patients with different expression levels of CK18 using randomized controlled study and provide evidence for the necessity of postoperative adjuvant TACE.

ELIGIBILITY:
Inclusion Criteria:

1. Via clinical diagnosis and confirm it is primary liver cancer
2. Pathological evidence of HCC
3. Estimate tumor can gain treatment of curing operation
4. No evidence for extrahepatic metestasis
5. liver function ：Child-Pugh A/B

Exclusion Criteria:

1. reject to attend；
2. impossible to come to our hospital for physical examination regularly.
3. cancer epitome、seed focus、lymph node or distant metastasis
4. Blood clotting function hindrance; 5, Patients with other diseases which may affect the treatment mentioned.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 320 patients with HCC
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2013-01; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 3 years

SECONDARY OUTCOMES:
Time to recurrence | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China